CLINICAL TRIAL: NCT05785156
Title: Diagnostic and Prognostic Value of New Quick Tests of Action Slowing in Stroke and in Cognitive Neurodegenerative Disease
Acronym: QTOAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0082
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Action Speed; Dementia Mild Cognitive Impairment; Alzheimer Disease
Keywords: executive processes; attention; Stroke; action speed; Diagnostic; sensitivity; specificity; dementia mild cognitive impairment; Alzheimer disease
MeSH Terms: conditions — Stroke; Alzheimer Disease; Disease; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute stroke patients
  Interventions: Other: quick tests
- cognitive neurodegenerative disorders: cognitive neurodegenerative disorders (Alzheimer Disease (AD), Lewy Body disease (LBD), FrontoTemporal lobar degeneration (FTLD), Cortico Basal Degeneration (CBD) and Progressive Supra Nuclear Palsy (PSNP)
  Interventions: Other: quick tests

INTERVENTIONS:
Other: quick tests — New quick tests are
  * Batterie MindPlus (Brevet n° FR1908081, Suarez 2019) is a quick reaction time battery and
  * Minimal Cognitive Evaluation (MCE) test (Sardi et al, 2019) is a cognitive screening tests including a specific assessment of slowing

SUMMARY:
A large series of recent studies have documented the frequency of the slowing of the action in brain diseases, especially vascular and neurodegenerative diseases. In stroke, the predictive value of action slowing at the acute phase for predicting post-stroke functional outcome remains poorly investigated. In neurodegenerative diseases, the diagnostic relevance of the slowing at the prodromal stage remains unknown and this diagnostic requires new tests. Finally, in terms of anatomical determinants, few studies have studied the determinants of action slowing. The objectives of this project are to Determine the diagnostic and prognostic value of action slowing assessed with new quick tests in patients with acute stroke (Neurovascular Unit) and cognitive neurodegenerative disorders (Alzheimer Disease (AD), Lewy Body disease (LBD), Fronto Temporal lobar degeneration (FTLD), Cortico Basal Degeneration (CBD) and Progressive Supra Nuclear Palsy (PSNP)) and to define the lesion determinants with VBM and VLSM

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40 and 85 years old,
* French native language,
* Social Security affiliation.
* University Memory Clinic for: Mild severity disorder (MMSE> 19) or major severity disorder related to AD : Albert 2011 criteria ; McKhann 2011
* to MCL according to McKeith criteria
* to FTLD according to Rascovsky 2011 criteria
* BBD according to Armstrong's criteria
* related to PSP according to Höglinger criteria

Exclusion Criteria:

* Mental retardation or guardianship
* Previously diagnosed dementia
* Other current or past brain condition
* severe head trauma
* epilepsy prior to stroke still requiring previous treatment
* Parkinson disease, multiple sclerosis...
* brain tumor or brain radiation therapy
* Current or past schizophrenia or psychosis
* Active or past psychiatric disorders requiring a stay> 2 days in a specialized environment
* Contra indication to MRI
* Comorbidity with life expectancy <1 year
* Comorbidity affecting cognition in particular:
* Alcohol (> 3 glasses / day) or history of alcohol withdrawal syndrome
* opiate or cocaine addiction or opiate withdrawal syndrome
* renal failure (dialysis or creatinine clearance <30)
* hepatic failure (spontaneous INR> 1.5 or PT <60%)
* respiratory failure requiring oxygen therapy
* heart failure (orthopnea> 2 pillows)
* persistent vigilance disturbances (NIHSS1a score ≤1)
* cancer with paraneoplastic syndrome
* treatment with gold salts, D Penicillamine or other treatment with cognitive effect
* Patient under guardianship or curators or private under public law
* Pregnant and / or lactating wom

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute stroke patients (Stroke Unit) and cognitive neurodegenerative disorder patients (Alzheimer Disease (AD), Lewy Body diseaese (LBD), FrontoTemporal lobar degeneration (FTLD), Cortico Basal Degeneration (CBD) and Progressive SupraNuclear Palsy (PSNP))
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Value of the speed of the action with the 'RT Componential Analysis of Action Speed' battery in all patients | 12 months
  RT Componential Analysis of Action Speed

SECONDARY OUTCOMES:
Speed values of action measured in all patients with the "MindPlus" battery in all patients | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No